CLINICAL TRIAL: NCT00427804
Title: Tumor Necrosis Factor-α Induces Vitamin D Resistance in Small Intestinal Calcium Absorption
Brief Title: Tumor Necrosis Factor Decreases Vitamin D Dependant Calcium Absorption
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Atlanta VA Medical Center (U.S. Federal Agency)
Collaborators: Emory University (Other)
Responsible Party: Principal Investigator, Vin Tangpricha, Staff Physician, Atlanta VA Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Vitamin D-2007
Record Dates: First submitted 2007-01-25; First posted 2007-01-29 (Estimated); Results first posted 2011-09-02 (Estimated); Last update posted 2013-02-04 (Estimated); Status verified 2013-01

CONDITIONS: Rheumatoid Arthritis; Crohn's Disease
Keywords: Calcium absorption; Vitamin D
MeSH Terms: conditions — Arthritis, Rheumatoid; Crohn Disease | interventions — Calcitriol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Calcitriol (Experimental): Calcitriol 0.25 mcg orally twice a day for 7 days or calcitriol 0.50 mcg orally twice a day for 7 days.
  Interventions: Drug: calcitriol

INTERVENTIONS:
Drug: calcitriol — 0.25 mcg PO BID for 1 week for low dose then 0.25 mcg PO BID for high dose

SUMMARY:
This study is a pilot study to determine whether patients with TNFα excess have decreased calcium absorption in response to calcitriol (1,25-dihydroxyvitamin D, the active form of vitamin D) compared to normal controls. This initial pilot study is being done to determine if it is feasible to conduct a study where TNFα could be blocked (e.g., by anti-TNFα therapy such as Enbrel® or Remicade®) to improve vitamin D dependant calcium absorption and thus bone health.

DETAILED DESCRIPTION:
Vitamin D is important for the maintenance of normal calcium homeostasis by improving the efficacy of calcium absorption from the small intestine. The efficacy of calcium absorption is decreased with aging, menopause, and other inflammatory states. Subjects who have low intestinal absorption of calcium are at risk for developing osteoporosis and fractures. Early data suggests that patients with rheumatoid arthritis (RA) and Crohn's disease appear to have decreased calcium absorption. Patients with RA and Crohn's disease have elevated levels of TNFα in local tissues and systemically which may be causing resistance to vitamin D dependant calcium absorption.

Recently a new vitamin D dependant calcium channel important for calcium absorption has been discovered in the small intestine called Transient Receptor Potential Vallinoid type 6 (TRPV6). We have some pre-clinical data in rats to suggest that TNFα has a role in inhibiting the expression of this protein by decreasing the induction of this protein in response to vitamin D treatment.

HYPOTHESIS:

Subjects with disease conditions that result in elevated TNFα have vitamin D resistance and inability to increase calcium absorption with increasing concentrations of calcitriol.

STUDY DESIGN:

Subjects: The study will be conducted at the Emory GCRC/Emory Clinic and VA clinical research center. Study participants will be recruited from the Atlanta Veterans Administration Medical Center (VAMC) and Emory Clinics for participation in the study according to the following inclusion and exclusion criteria

Inclusion: Males, age 18 to 50, history of Crohn's disease or Rheumatoid Arthritis (cases) or healthy individuals (controls)

Exclusion: Subjects already taking activated vitamin D medications such as calcitriol, Zemplar®, Hectoral®, vitamin D deficiency defined as 25(OH)D ≤ 20 ng/ml, post-menopausal women (absence of menses for greater than 6 months by history or FSH level >20), history of nephrolithiasis, history of hypercalcemia or hypercalciuria, short bowel disease, glucocorticoid use, use of osteoporosis medication (bisphosphonate, calcitonin or teriparatide), chronic kidney disease (calculated GFR <60 ml/min/1.73 m2), history of hyperparathyroidism (PTH greater than upper limit of normal) or hypoparathyroidism (PTH below lower limit of normal)

Procedures:

Screening Phase: Case subjects will be identified from Rheumatology and Gastroenterology clinics from the VA or Emory Clinic. The subject's doctors will give the patient a brochure of the study with the study investigator's name and phone number to contact. There will also be advertisements in the Rheumatology and Gastroenterology clinics to recruit subjects for the study. Control subjects will be identified by postings at the VA hospital or at Emory Clinic in designated areas for research postings.

The subject will initiate contact with the study personnel by calling the number on the advertisement or brochure. The study investigator will pre-screen the subject on the phone to see if the subject is eligible for entry into the study. If the subject remains eligible, the subject will be invited to the VA clinical research center or Emory GCRC/Emory Clinic for informed consent.

Screening Visit: The study investigator will review the inclusion and exclusion criteria with each subject. If the subject agrees to participate in the study, the subject will sign the informed consent and undergo baseline laboratory investigations for total calcium, parathyroid hormone (PTH), 25-hydroxyvitamin D, comprehensive panel including renal function, 24-hour urine collection for calcium and creatinine clearance. Subjects will be counseled to take no more than 600 mg of calcium daily and no more than 400 IU a day of vitamin D. The subjects will be instructed on how to complete a three day food diary for future visits.

They will be given a schedule to return for the following visits.

Visit #1 (baseline fractional absorption of calcium (FCA)) Subjects will return to the clinical research center in a fasting state for a baseline FCA test (see specific methods in the following section). Subjects will return their three day food diary record. Subjects will also have blood drawn for comprehensive panel including calcium and renal function, 1,25-dihydroxyvitamin D, PTH level and serum TNFα. The subjects will be given calcitriol 0.25 mcg PO BID to be taken for 7 days.

Visit #2 (FCA on low dose calcitrol, 0.25 mcg PO BID) Subjects will take their morning dose of calcitriol 8 am on the day of visit #2. Subjects will come to the clinic in a fasting state. They will return their 3 day food diary records. A repeat FCA will be performed. Subjects will also have blood drawn for comprehensive panel including calcium and renal function, 1,25-dihydroxyvitamin D, PTH level and serum TNFα. After the test is completed, the subjects will be given calcitriol 0.50 mcg PO BID to be taken for 7 days. They will be scheduled to return to the clinical research center within 20 days after a minimum 7 day washout period.

Visit #3 (FCA on high dose calcitriol, 0.50 mcg PO BID) Subjects will take their morning dose of calcitriol at 8 am on the day of visit #3. Subjects will come to the clinic in a fasting state. They will return their 3 day food diary records. A repeat FCA will be performed. Subjects will also have blood drawn for comprehensive panel including calcium and renal function, 1,25-dihydroxyvitamin D, PTH level and serum TNFα.

Fractional absorption of calcium (FCA) procedure Subjects will come to the clinic after an overnight fast. After voiding the fasting urine, a 24 hour urine collection will begin. Each subject will receive a standard breakfast (see FCA diet section) which will contain approximately 211 mg of calcium and 45 IU of vitamin D. Oral 43Ca will be administered after the patient has drunk the milk. 1.9 ml will be drawn from a sterile 43Ca (calcium chloride) vial with a syringe and will be injected in 4 ounces of distilled water. The subject will drink the glass of water. The glass will be rinsed twice with 4 ounces of distilled water and the subject will drink each rinse.

2.7 ml of 42Ca will be drawn from a sterile 42Ca (calcium chloride) vial with a sterile hypodermic syringe. The solution will be injected into the patient intravenously with an IV catheter and flushed with 5 ml of normal saline. The intravenous calcium will be infused within 30 minutes of ingestion of the oral calcium.

The subject will be discharged from the clinical research center and will continue with their 24 hour urine collection. The following morning, the subject will return the 24 hour urine collection to the research clinic. The subject will be advised to not eat for at least 4 hours after the breakfast meal.

ELIGIBILITY:
Inclusion Criteria:

* Males
* Age 18 to 50
* History of Crohn's disease or Rheumatoid Arthritis (cases) or healthy individuals (controls)

Exclusion Criteria:

* Subjects already taking activated vitamin D medications such as calcitriol, Zemplar®, Hectoral®
* Vitamin D deficiency defined as 25(OH)D ≤ 20 ng/ml
* Post-menopausal women (absence of menses for greater than 6 months by history or FSH level >20)
* History of nephrolithiasis
* History of hypercalcemia or hypercalciuria
* Short bowel disease
* Glucocorticoid use
* Use of osteoporosis medication (bisphosphonate, calcitonin or teriparatide)
* Chronic kidney disease (calculated GFR <60 ml/min/1.73 m2)
* History of hyperparathyroidism (PTH greater than upper limit of normal) or
* Hypoparathyroidism (PTH below lower limit of normal)

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2007-01; Primary Completion 2009-08 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vin Tangpricha, M.D. Ph.D., Principal Investigator — Emory University
Locations (1):
- Atlanta VAMC, Atlanta, Georgia, United States

REFERENCES:
- [Result] Kumari M, Khazai NB, Ziegler TR, Nanes MS, Abrams SA, Tangpricha V. Vitamin D-mediated calcium absorption in patients with clinically stable Crohn's disease: a pilot study. Mol Nutr Food Res. 2010 Aug;54(8):1085-91. doi: 10.1002/mnfr.200900351. PMID 20306476

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was conducted July 2007 to August 2008 at the Atlanta VA Medical Center.
Pre-assignment Details: Subjects included those with Crohn's disease and healthy controls.
Groups:
- Crohn's Disease: Subjects with stable Crohn's disease
Period: Overall Study
Arm/Group | Healthy Control | Crohn's Disease
Started | 4 | 5
Completed | 4 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Healthy Control | Crohn's Disease | Total
Number analyzed (Participants) | 4 | 5 | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 5 | 9
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 42.40 (5) | 35.5 (10) | 39.3 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 4 | 5 | 9
Region of Enrollment [Number; unit: participants]
  United States | 4 | 5 | 9

OUTCOME MEASURES:

1. Primary Outcome: Intestinal Absorption of Calcium
Time Frame: 12 Weeks
Reporting Status: Not Posted

2. Primary Outcome: Fractional Absorption of Calcium
Description: Fractional absorption of calcium (see citation for complete details)
Time Frame: 7 week
Measure: Number; unit: Percentage of absorption
Arm/Group | Healthy Control | Crohn's Disease
Number analyzed (Participants) | 4 | 5
Percentage of absorption | 71 | 115

ADVERSE EVENTS:
Arm/Group | Healthy Control | Crohn's Disease
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/5
Other Adverse Events (participants affected / at risk) | 0/4 | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No